CLINICAL TRIAL: NCT01209273
Title: Prospective, Observational and Multi-center Study of a Comparison of Quality of Life on Automated Peritoneal Dialysis and Continuous Ambulatory Peritoneal Dialysis
Brief Title: Comparison of Quality of Life on Automated Peritoneal Dialysis and Continuous Ambulatory Peritoneal Dialysis
Acronym: EQlips
Status: Completed | Type: Observational
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: Clinical Research Center for End Stage Renal Disease, Korea (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Yong-Lim Kim, Professor, Kyungpook National University Hospital
Other Study IDs: A-01
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2015-09-15 (Estimated); Status verified 2015-09

CONDITIONS: End Stage Renal Disease; Peritoneal Dialysis
Keywords: Quality of Life; Automated Peritoneal Dialysis; Continuous Ambulatory Peritoneal Dialysis; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood 24hr urine PD dialysate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- APD group: which can be 3 to 5 exchanges daily, and up to 20 liters daily( including up to two daytime exchanges)
- CAPD group: which can be 1 to 4 exchanges daily and up to 16 liters daily(including up to two daytime exchanges)

SUMMARY:
The objective of this study is to compare Quality of Life (QoL) between Automated Peritoneal Dialysis (APD) and Continuous Ambulatory Peritoneal Dialysis (CAPD).

DETAILED DESCRIPTION:
Automated peritoneal dialysis (APD) was first described in 1981, 5 years after the introduction of continuous ambulatory peritoneal dialysis (CAPD). It is increasingly used increasingly used in comparison with CAPD from 20% in 1995 to more than 33% of PD patients in North America in 1998, and in 2000, 54% of PD patients in the United States performed some form of APD.

APD has been several advantages over CAPD such as reduced incidence of peritonitis, mechanical complications and greater psychosocial acceptability. Many studies demonstrated a benefit for APD. In one Mexican retrospective study, APD has a better technical survival than CAPD with improvement of 1st peritonitis episode and French registry data showed the better peritonitis-free probability and autonomy in APD compared to CAPD. One study found that peritonitis rates and hospitalization were significantly less in patients on APD when results were expressed as episode/patient-year. Also a small randomized clinical trial comparing APD and CAPD showed that APD can help to keep selected patients vocationally or socially active.

Although APD has been expected to improve better condition of peritoneal dialysis patients, convincing evidence of major advantages is lacking and a benefit for APD is not demonstrated.

In three of randomized clinical trials, APD, APD did not differ from CAPD with respect to mortality (RR 1.49, 95% CI 0.51 to 4.37), risk of peritonitis(RR 0.75, 95% CI 0.50 to 1.11), switching from original PD modality to a different dialysis modality(RR 0.50, 95% CI 0.25 to 1.02), hernias(RR 1.26, 95% CI 0.32 to 5.01), PD fluid leaks(RR 1.06, 95% CI 0.11 to 9.83), PD catheter removal ( RR 0.64, 95% CI 0.27 to 1.48) or hospital admissions (RR0.96, 95% CI 0.43 to 2.17). In addition APD has potential disadvantages compared with CAPD like a possible faster in residual renal function, less sodium removal and more peritoneal protein loss and more expensive than CAPD. All of three large cohorts, NECOSAD, USRDS and ANZDATA showed that the risk of technical failure was not different between APD and CAPD but similar.

Because results on comparison between APD and CAPD is vague, prospective, observational and multi-center study in incident patients are required to gain more insight into survival on APD compared with CAPD in the course of peritoneal dialysis.

Quality of Life is an important outcome parameter when advising patients on renal replace treatment modality section. The introduction of a machine to assist the patient with PD exchanges can potentially improve quality of life in different ways. De Wit et al. analyzed health-related quality of life (HRQOL) in 37 APD and 59 CAPD patients from 16 different Dutch dialysis centers. In a multivariate analysis, the mental health was found to be better in APD as compared to CAPD patients. In addition, there were indications that APD patient tended to be less depressed and anxious than CAPD patients. In a prospective randomized trial, Bro et al. found no difference between CAPD and APD patients in quality of life measures. However APD patient tended to have more time for work, family, and social activities as compared to CAPD patients.

From these limited data, it can possibly be concluded that quality of life is very important to evaluate the lifestyle of the patient and to adapt the PD regimen.

Therefore, quality of life (QoL) assessment is expected to evidence to support the hypothesis that APD is superior to CAPD.

And the incidences of clinical events treatment modality change, peritonitis episode, exit site/tunnel infection, hospitalization, death, cancer development) are also reviewed to support that hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects at least 20 and older at that time of obtaining informed consent
* Subjects performing CAPD or APD
* Subject with a total Kt/V≥ 1.7 at baseline

Exclusion Criteria:

* Subjects who have undergone abdominal surgery within the last 30 days except for PD catheter insertion
* Subjects who is planned for renal transplantation or hemodialysis within 1 year following the date of informed consent
* Subjects who have received antibiotics for the treatment of peritonitis, exit-site or tunnel infection within the last 30 days
* Subjects who have active liver disease such as cirrhosis of the liver, active hepatitis or other active liver disease as evidenced by biopsy, laboratory (unstable liver enzymes over the last 90 days) or clinical examination.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Incident PD patients in Korea
Sampling Method: Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change in Quality of Life | 1yr
  change in quality of life and patient satisfaction scores from start to dialysis to 1yr between APD group and CAPD group.

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Lim Kim, M.D., Ph.D., Principal Investigator — Division of Nephrology, Department of Internal Medicine, Kyungpook National University School of Medicine
Locations (11):
- South Korea (11):
  - Inje University Haeundae Paik Hospital, Busan
  - Samsung Changwon Hospital, Changwon
  - Chungbuk National University Hospital, Cheongju-si
  - Kyungpook National University Hospital, Daegu
  - Daegu Fatima Hospital, Daegu
  - Eulji University Hospital, Daejeon
  - Chosun University Hospital, Gwangju
  - Jeju National University Hospital, Jeju City
  - Korea University Anam Hospital, Seoul
  - Eulji General Hospital, Seoul
  - St. Carolo Hospital, Suncheon